CLINICAL TRIAL: NCT02975544
Title: Pilot Study of CRECES Programme: Promoting Healthy Life Styles in Children Through the Social and Emotional Competence
Brief Title: An Exploratory Trial of a Health Education Programme Based on the Social and Emotional Competence in Children
Acronym: CRECES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Fundación Caja Navarra (Unknown)
Responsible Party: Principal Investigator, Elena Bermejo, Principal Investigator, Clinica Universidad de Navarra, Universidad de Navarra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 70801
Record Dates: First submitted 2016-11-15; First posted 2016-11-29 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Health Behavior; Emotional Intelligence
Keywords: social and emotional competence; healthy lifestyles; children; educational programme
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Received CRECES programme during 5 weeks as part of the extracurricular plan
  Interventions: Behavioral: CRECES programme
- Control group (No Intervention): Continued with their habitual school routine

INTERVENTIONS:
Behavioral: CRECES programme — The first unit of CRECES programme was implemented in 8 sessions. Each session was 40-50 minutes long and delivered during four weeks. Parents were provided with home-extension activities.
  Arms: Intervention group

SUMMARY:
The purpose of this study was to evaluate whether an intervention based on the social and emotional competence development improves the healthy lifestyles adoption in young children.

DETAILED DESCRIPTION:
This study has designed, implemented and evaluated an intervention to promote healthy lifestyles in children addressing the development of the social and emotional competence. This research followed the first three stages of the Medical Research Council framework for complex interventions: the theoretical, modeling phase and the exploratory trial. A randomised control trial with 37 children (5 y 6 years old) was conducted at the exploratory trial. The first unit was implemented in 8 sessions. A multi-method and multi-informant approach was used to assess the preliminary efficacy, acceptability and feasibility of the programme.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5 and 6 enrolled in a public school in the north of Spain

Exclusion Criteria:

* Children with severe cognitive or language special needs

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2015-03; Primary Completion 2015-04 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Changes on children's emotional knowledge | Baseline; Post-test (1 month), 7 months follow-up
  Directly measured on children by PERCEVAL test (Mestre, J. M., Guil, R., Martínez-Cabañas, F., Escandón, C. L., y Gonzalez de la Torre, G. (2011).

SECONDARY OUTCOMES:
Changes on the total and parcial dimensions (cooperation, independence and interaction) of children's basic social skills | Baseline, post-test (1 month) and 7 months follow-up
  Reported by parents by Preschool and Kindergarten Behavior Scales (PKBS-II; Merrell, 2003).
Changes on the total and parcial dimensions (comfort, satisfaction, resilience, risk avoidance and achievement) of children's health profile | Baseline, post-test (1 month) and 7 months follow-up
  Reported by children and parents by Child Health and Illness Profile-CHILDREN Edition (CHIP-CE; Rajmil, L., Serra-Sutton, V., Alonso, J., Herdman, M., Riley, A., y Starfield, B. (2003)

OTHER OUTCOMES:
Acceptability of the programme by children and parents who took part in | post-test (1 month)
  Explored by semi-structured interviews with children and parents
Efficacy on children social and emotional skills and healthy habits adoption perceived by parents | post-test (1 month)
  Explored by semi-structured interviews with parents
Feasibility of the programme's implementation | Baseline
  Examined by researcher's field diary

CONTACTS AND LOCATIONS:
Overall Officials: Elena Bermejo Martins, Nursing, PhD, Principal Investigator — University of Navarra

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bermejo-Martins E, Mujika A, Iriarte A, Pumar-Mendez MJ, Belintxon M, Ruiz-Zaldibar C, Lopez-Dicastillo O. Social and emotional competence as key element to improve healthy lifestyles in children: A randomized controlled trial. J Adv Nurs. 2019 Aug;75(8):1764-1781. doi: 10.1111/jan.14024. Epub 2019 Jul 8. PMID 30972808